CLINICAL TRIAL: NCT04180176
Title: A Multicenter, Low-Interventional Study to Evaluate the Feasibility of a Prospective Clinicogenomic Program
Brief Title: Prospective Clinicogenomic Program
Acronym: PCG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Flatiron Health, Inc.; Foundation Medicine, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GX41563
Record Dates: First submitted 2019-11-19; First posted 2019-11-27 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC); Small-Cell Lung Cancer (SCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- All-Comer Cohort (Experimental): Participants with mNSCLC or ES-SCLC will give blood samples at three separate timepoints for ctDNA profiling.
  Interventions: Other: Blood Draw
- Front-line Immunotherapy Re-enrollment Cohort (Experimental): Participants with mNSCLC or ES-SCLC that have received front-line treatment as defined by the protocol will give blood samples at three separate timepoints for ctDNA profiling.
  Interventions: Other: Blood Draw

INTERVENTIONS:
Other: Blood Draw — Participants will have blood drawn at enrollment, the first tumor assessment, and at disease progression or end of therapy.

SUMMARY:
The main purpose of this study is to evaluate the feasibility of a scalable, prospective research program for participants with metastatic non-small cell lung cancer (mNSCLC) or extensive-stage small-cell lung cancer (ES-SCLC) planning to start standard-of-care (SOC) systemic anti-cancer treatment. The study will also examine ctDNA status over the course of treatment as a predictor of response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of mNSCLC or ES-SCLC
* Planned initiation of SOC systemic anti-cancer treatment
* Front-Line Immunotherapy Cohort: Received front-line treatment of an immune blockade therapy including anti-CTLA-4, anti-PD-1, or anti-PD-L1 therapeutic antibody on Protocol GX41563

Exclusion Criteria:

- Participant actively receiving investigational medicinal product(s) as part of an interventional trial at the time of signing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 945 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Proportion of Potential Eligible Participant Enrollment | Up to 5 years
Proportion of Enrolled Participants Submitting Sufficient Blood Samples | At enrollment, then at pre-defined intervals from the first tumor assessment until disease assessment or end of therapy, whichever comes first, for up to 5 years.

SECONDARY OUTCOMES:
Blood Level of ctDNA | At enrollment, then at pre-defined intervals from the first tumor assessment until disease assessment or end of therapy, whichever comes first, for up to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- United States (23):
  - Alabama Oncology, Birmingham, Alabama
  - Clearview Cancer Institute, Huntsville, Alabama
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Yale University, New Haven, Connecticut
  - Florida Cancer Specialists; Department of Oncology, Fort Myers, Florida
  - Florida Cancer Specialist, North Region, St. Petersburg, Florida
  - SCRI Florida Cancer Specialists PAN, Tallahassee, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - University Cancer & Blood Center, LLC; Research, Athens, Georgia
  - Piedmont Cancer Institute, PC, Atlanta, Georgia
  - Fort Wayne Med Oncology & Hematology Inc, Fort Wayne, Indiana
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Jackson Oncology Associates, PLLC, Jackson, Mississippi
  - Southeast Nebraska Cancer Ctr, Lincoln, Nebraska
  - Regional Cancer Care Associates LLC, Central Jersey Division, East Brunswick, New Jersey
  - Hematology Oncology Associates of Central New York, East Syracuse, New York
  - West Clinic, New York, New York
  - National Translational Research Group, Port Jefferson Station, New York
  - Oklahoma Cancer Specialists and Research Institute, Tulsa, Oklahoma
  - SCRI Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Hematology Oncology Associates of Fredericksburg, Inc., Fredericksburg, Virginia
  - Virginia Cancer Institute - Richmond, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).